CLINICAL TRIAL: NCT07277699
Title: Effects of Otago and Frenkel's Exercises on Strengthening of Antigravity Muscles in Parkinson's Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0051; uol (Other: UOL/IREB/25/09/0051)
Record Dates: First submitted 2025-08-26; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-08

CONDITIONS: Parkinson
Keywords: Otago,Frenkel's exercises,Parkinson's

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Otago Exercise Program (Experimental): 20 Participants in this arm will undergo a combined exercise program consisting of the Otago Exercise Program (OEP) and conventional Physiotherapy. The intervention is designed to strengthen antigravity muscles (hip, knee, and trunk extensors), improve balance, coordination, and functional mobility, and reduce fall risk in patients with Parkinson's disease.
  Interventions: Behavioral: Otago exercises
- Frenkel's Exercise Program (Experimental): 20 Participants in this arm will under go Frenkel's Exercises program and conventional physiotherapy. This intervention help Parkinsons patient by improving coordination, balance and enhance motor learning and confidence
  Interventions: Behavioral: Frenkels exercise

INTERVENTIONS:
Behavioral: Otago exercises — After collecting the patient's data appropriate modalities will be applied to initiate the treatment session. This includes the use of an Electric Heating pad on the lower limb for 10 mints. Gentle walking will be performed for 1 mints along with arm swing (10 repetitions) and neck stretching focusing on upper trapezius muscle (3 repetition).After that the12 steps of Otago exercise will be performed with 10 repetition.Total session time is 40 mints.
  Arms: Otago Exercise Program
Behavioral: Frenkels exercise — After collecting the patient's data sessions will be delivered 3 times per week lasting for 40 mints only and than appropriate modalities will be applied to initiate the treatment session. This includes the use of an Electric Heating pad on the lower limb for 10 mints. Gentle walking will be performed for 1 mints along with arm swing (10 repetitions) and neck stretching focusing on upper trapezius muscle (3 repetition).After that the steps of Frenkels exercise program will be performed on patients with 10 repetition.
  Arms: Frenkel's Exercise Program

SUMMARY:
Using both Otago and Frenkel's exercises offers complementary benefits building muscle strength and refining coordination in anti-gravity muscles making daily activities safer and more fluid for people with Parkinson's.

DETAILED DESCRIPTION:
Combining Otago and Frenkel's exercises can slow functional decline, reduce falls, and improve quality of life for Parkinson's patients. These programs empower patients and families by promoting active participation in care rather than relying only on medications. Early introduction, guided by physiotherapists, gives the best outcomes helping patients stay mobile, confident, and independent for longer.

ELIGIBILITY:
Inclusion Criteria:

1. Patient diagnosed with parkinsons disease using the Hoehn and Yahr scale
2. Patient age 55-75.
3. Both male and female.
4. Able to walk independently.
5. Willing and ability to provide information consent to participate in study. -

Exclusion Criteria:

1. Presence of other neurological condition(stroke, multiple sclerosis).
2. severe cardiovascular disease.
3. major psychiatric disorder.
4. currently participating in other study.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-08-18 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Antigravity muscle strenght (Manual Muscle strength). | Baseline before treatment (week 0) post -interventiom (week 4 )
  Strength of major antigravity muscle including Hip muscles, Knee muscles and ankle muscles.
  strength evaluated by using Manual Muscle Testing based on oxford Grading Scale (0-5).
  . Grade 0 ( No contraction).
  * Grade 1 (trace): slightly contraction detected but no movement occur at joint.
  * Grade 2 (poor): Full range of motion in a gravity eliminated position.
  * Grade 3(Fair): Full range of motion against gravity.
  * Grade4 (Good): Full range of motion against gravity moderate resistance.
  * Grade5 (Normal) Full Range of motion against gravity and maximum resistance. Participants tested in standardized position for each group. unit of measurement : MMT grade (0-5)
Balance and reduction in fall risk. | baseline Before treatment (0 Week) post- intervention ( 4 week )
  Balance assessed through the Berg Balance Scale (BBS). Berg Balance Scale items: 14 Tasks (sit to stand, standing, stepping, unsupported, reaching, turning) total score (0-56) scoring:0-4 for each task Maximum score=56 41-56=low Fall risk 21-40=Medium Fall risk 0-20=High Fall risk

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lahore, Gujranwala, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No